CLINICAL TRIAL: NCT03076866
Title: Suivi Prospectif Des Patients Presentant un Rhumatisme Inflammatoire Chronique
Brief Title: Prospective Follow-up of Patients With Chronic Inflammatory Rheumatism
Acronym: PPCRNice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Principal Investigator, Service de Rhumatologie, Professor, Centre Hospitalier Universitaire de Nice
Other Study IDs: 260
Record Dates: First submitted 2017-02-23; First posted 2017-03-10 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Inflammatory Disease; Rheumatoid Arthritis; Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational follow-up:clinical, radiological et biological

SUMMARY:
It is a prospective follow-up. The aim is to study the maintenance of therapeutic at 10 years and 20 years of inflammatory rheumatism (rheumatoid arthritis and spondyloarthritis)

DETAILED DESCRIPTION:
All subjects were followed up on a yearly basis collection with clinical data (weight, sex, age, comorbidities, treatment), biological (VS, CRP, ACPA, lipid balance, cross laps), radiology (hand and foot radiographs and ultrasonography ), BMO Measure

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years
* Rheumatoid arthritis meeting ACR criteria Spondyloarthritis meeting ASAS criteria

Exclusion Criteria:

* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patients with a inflammatory disease (rheumatoid arthritis and spondyloarthritis) follow-up in the rheumatologic department
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2001-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
therapeutic maintenance at 20 years of follow-up | 20 years
  All subjects benefit from an annual follow-up including a collection of clinical data (age, sex, weight, comorbidities, swelling and painful joints), biological (CRP, ACPA, cross laps, lipids), radiological, BMO measures (Hologic), and treatments (biological and synthetic DMARDS). Each rheumatologic modification or stop of treatment is transcribed. Therapeutic maintenance definition: modification in rheumatologic treatment (number of DMARDS at 20 years)

SECONDARY OUTCOMES:
evolution of lipidics parameters at 20 years of follow-up | 20 years
  lipidics parameters ( total, HDL, LDL cholesterol and tryglicerides) are collected each years and modifications/evolution of these parameters will be studied

OTHER OUTCOMES:
evolution of BMD at 20 years of follow-up | 20 years
  each 2 years during visit of follow up, BMD parameters (Hologic QDR 4500A measurements performed in pasteur 2 hospital: tscore, Zscore and BMD in in g/cm2) are collected. Osteopenia was defined by a T-score between -1 and -2.5 SD and osteoporosis by a T-score below -2.5 SD, in accordance with the World Health Organization guidelines. evolution of BMD will be studied in relation with rheumatologics treatments

CONTACTS AND LOCATIONS:
Overall Officials: christian roux, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- rheumatology department CHU nice, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided